CLINICAL TRIAL: NCT04243629
Title: Co-administration of Pramlintide and Insulin Via an Automated Dual-hormone Artificial Pancreas System to Regulate Glucose Levels in Adults Living With Type 1 Diabetes: a Randomized, Controlled, Crossover Trial.
Brief Title: Co-administration of Pramlintide and Insulin Via an Automated Dual-hormone Artificial Pancreas System in Adults With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020-6258
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 1; Type 1 Diabetes; Postprandial Hyperglycemia
Keywords: Artificial pancreas; Closed-loop system; Amylin; Pramlintide; Type 1 Diabetes; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia | interventions — Insulin, Short-Acting; pramlintide; Pancreas, Artificial

STUDY DESIGN:
Intervention Model Description: This is a two-way, randomized, open-label, controlled, crossover trial to compare the following strategies:
  (i) Rapid insulin-plus-Pramlintide closed-loop delivery
  (ii) Rapid insulin-plus-Placebo closed-loop delivery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid Insulin-Plus-Pramlintide (Experimental): Rapid insulin and pramlintide infusion in two insulin pumps
  Interventions: Drug: Rapid-Acting Insulin; Drug: Pramlintide Acetate; Device: Artificial Pancreas
- Rapid Insulin-Plus-Placebo (Placebo Comparator): Rapid insulin and placebo (saline) infusion in two insulin pumps
  Interventions: Drug: Rapid-Acting Insulin; Drug: Placebo; Device: Artificial Pancreas

INTERVENTIONS:
Drug: Rapid-Acting Insulin — Novorapid or Humalog insulin delivered in a basal-bolus manner.
Drug: Placebo — Placebo (saline) delivered in a basal-bolus manner at a fixed ratio with insulin.
  Arms: Rapid Insulin-Plus-Placebo
Drug: Pramlintide Acetate — Pramlintide acetate delivered in a basal-bolus manner at a fixed ratio with insulin.
  Arms: Rapid Insulin-Plus-Pramlintide
Device: Artificial Pancreas — Tandem insulin pump, Dexcom G6 sensor, study smartphone running the iMAP algorithm.

SUMMARY:
One of the main challenges in maintaining tight glucose control in a closed-loop system occurs at meal times. Amylin is a gluco-regulatory beta-cell hormone that is co-secreted with insulin in response to nutrient stimuli, and is deficient in patients with type 1 diabetes. Amylin, in the postprandial period, contributes to regulating glucose levels by delaying gastric emptying, suppressing nutrient-stimulated glucagon secretion, and increasing satiety. Pramlintide is a synthetic analog of the hormone amylin. A closed-loop system that delivers both insulin and pramlintide, based on glucose sensor readings, has the potential to better normalize glucose levels, especially during the post-prandial period.

The aim of this project is to assess whether co-administration of pramlintide with rapid insulin in an artificial pancreas system will improve glycemic control in adults with Type 1 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent
2. Males and females ≥ 18 years of age
3. HbA1c ≤ 11% (this is so we also include patient that are potentially missing some meal boluses)
4. Insulin pump use for at least 6 months and actively performing carbohydrate counting
5. Clinical diagnosis of type 1 diabetes for at least 12 months. The diagnosis of T1D is based on the investigator's clinical judgment; C peptide level and antibody determinations are not planned.
6. Women of child-bearing potential must be ready and able to use a highly effective method of birth control. Women of childbearing potential are females who have experienced [the first occurrence of menstruation] and do not meet the criteria for women not of childbearing potential. Women not of childbearing potential are females who are permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.

Exclusion Criteria:

1. Current total daily dose < 0.4 units/kg (we wish to exclude participants who would still be considered in honeymoon period).
2. Current or ≤ 1 month use of other antihyperglycemic agents (SGLT2 inhibitors, GLP-1 agonists, Metformin, Acarbose, etc.…).
3. Current use of glucocorticoid medication (except low stable dose and inhaled steroids).
4. Anticipated need to use acetaminophen during study participation
5. Use of medication that alters gastrointestinal motility.
6. Planned or ongoing pregnancy.
7. Breastfeeding individuals.
8. Severe hypoglycemic episode within 3 months of admission.
9. Severe diabetes ketoacidosis episode within 3 months of admission.
10. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
11. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
12. Known hypersensitivity to any of the study drugs or their excipients.
13. Individuals with confirmed gastroparesis.
14. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
15. In the opinion of the investigator, a participant who is unable or unwilling to observe the contraindications of the study devices.
16. Unable to travel to research center within 3h if needed during study interventions
17. Failure to comply with team's recommendations (e.g. not willing to eat meals/snacks, not willing to change pump parameters, etc.).

Discontinuation Criteria:

1. Failure to comply with the protocol.
2. Pregnancy.
3. After an event which the PI believes it is not in the best interest for the patient to continue the trial.
4. The subject wants to withdraw consent to participate
5. The subject needs to take any medications that are contraindicated in the study
6. The subject can no longer be treated with the study medication for other reasons
7. The subject experiences severe hypoglycaemia requiring hospitalization or repeated hypoglycaemia requiring assistance to treat.
8. The subject fails to follow instructions given about the trial
9. The Study Team has decided to discontinue or terminate the clinical trial prematurely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Time in target range | 4 weeks
  Time each participant spent with glucose level in target range (3.9 - 10.0 mmol/L)

SECONDARY OUTCOMES:
Time between 3.9 - 7.8 mmol/L | 4 weeks
  Percentage of time each participant spent with glucose levels between 3.9 - 7.8 mmol/L
Time below 3,9, 3.3, and 2.8 mmol/L | 4 weeks
  Percentage of time each participant spent with glucose levels below 3.9, 3.3, and 2.8 mmol/L
Time above 7.8, 10.0, 13.9, 16.7 mmol/L | 4 weeks
  Percentage of time each participant spent with glucose levels above 7.8, 10.0, 13.9, and 16.7 mmol/L
Mean glucose level | 4 weeks
  Each participant's mean glucose level
Total insulin delivery | 4 weeks
  Each participant's total insulin delivery
Standard deviation and coefficient of variance | 4 weeks
  Each participant's standard deviation and coefficient of variance of glucose levels as a measure of glucose variability
Gastrointestinal symptoms | 4 weeks
  Number of each participant's gastrointestinal symptoms
Number of hypoglycemia events | 4 weeks
  Each participant's number of hypoglycemia events defined as at least 15 min below 3.0 mmol/L with the end of the event being 15 minutes > 3.9 mmol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The raw data (i.e., insulin delivery, glucose levels, individual participant data) and informed consent form could be shared by the corresponding author, ahmad.haidar@mcgill.ca, upon reasonable request for academic purposes, subject to Material Transfer Agreement and approval of McGill University Health Center's Research Ethics Board. All data shared will be deidentified. Study protocol is available with publication.
Supporting Information: Study Protocol, ICF